CLINICAL TRIAL: NCT04603482
Title: Self-Management Interventions: Considering Needs & Preferences of Dementia Caregivers
Brief Title: Self-Management Intervention: Considering Needs & Preferences of Dementia Caregivers (Caregiver Career Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Jaclene A. Zauszniewski, Principal Investigator, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01NR018476 (NIH)
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Stress; Carer Stress Syndrome; Dementia; Alzheimer's Disease; Bereavement
Keywords: Caregiver; Biofeedback; Resourcefulness; Self-Management
MeSH Terms: conditions — Dementia; Alzheimer Disease | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants were aware of which intervention they were receiving (Resourcefulness Training, HRV-focused BioFeedback, Attention Control: Diversonal Activities, but were not aware of which arm they had been randomly assigned to, or whether their intervention was an active or placebo comparator. The PI and Outcomes Assessor were blinded as to the identity of individual participants, and, during data collection, which participants had been assigned to which arm/intervention. In order to complete study aims, variables indicating arm and intervention assignment were included in the final data file.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-management intervention based on Need (Active Comparator): Participants randomly assigned to this arm receive a self-management intervention (Resourcefulness Training or Biofeedback) according to baseline data.
  Interventions: Behavioral: Resourcefulness training; Behavioral: Biofeedback
- Self-management intervention based on Preference (Active Comparator): Participants randomly assigned to this arm receive a self-management intervention (Resourcefulness Training or Biofeedback) according to their preference.
  Interventions: Behavioral: Resourcefulness training; Behavioral: Biofeedback
- Attention Control: Diversonal Activities (Placebo Comparator): Participants randomly assigned to this arm will be presented with diversional activities.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Resourcefulness training — Resourcefulness training is a cognitive behavioral intervention that consists of teaching and reinforcing personal (self-help) and social (help-seeking) strategies to overcome adversity.
  Arms: Self-management intervention based on Need; Self-management intervention based on Preference
Behavioral: Biofeedback — Biofeedback training combines teaching slow, deep, paced breathing with real-time tracking to increase an individual's heart rate variability and ultimately improve self-regulation.
  Arms: Self-management intervention based on Need; Self-management intervention based on Preference
Behavioral: Attention Control — Participants randomly assigned to this intervention will receive suggested Diversional Activities, presented in an audiovisual format.
  Arms: Attention Control: Diversonal Activities

SUMMARY:
How do varying levels of participation in selecting self-management interventions (ranging from no input into the selection to selection based on need or preference) affect health risks and physical and mental health over time in family caregivers of persons with Alzheimer's and other dementia disorders? Caregivers will be randomized to 1) information on diversional activities (attention control); 2) self-management intervention based on need (SM-need); or 3) self-management intervention of their preference (SM-preference).

DETAILED DESCRIPTION:
The study has two aims: The primary aim (A1) is to examine differences across the three groups (attention control, SM-need, and SM-preference) on caregiver health (health risks and mental and physical health) over time. The investigators hypothesize that the caregivers who receive a self-management intervention based on need (SM-need) or preference (SM-preference) will have better health outcomes than those in the attention control.

Secondary aims are to: A2) explore whether caregiver baseline need or preference for intervention (i.e. choice) is associated with: a) care recipient's symptoms; b) caregiver reactions; and c) caregiving involvement, and A3) build caregiver profiles from demographic/ contextual factors that are associated with their needs and preferences for the self-management interventions.

All caregivers will complete assessment measures and measures of health risks, and physical and mental health at baseline (T1), about 6 months (T2), and about 12 months (T3). Caregivers will be randomly assigned to one of three groups. The attention control group will receive information on diversional activities. The SM-need group will receive a self-management intervention for biofeedback training or resourcefulness training, as determined by baseline cut scores. Caregivers in the SM-preference group will choose one of the two self-management interventions according to their personal preference.

Both self-management interventions (biofeedback training, resourcefulness training) and the diversional activities, are delivered over four weeks (between T1 and T2). Caregivers may use the intervention whenever and as often as they wish (i.e. self-tailoring) for the remainder of the study period. These resourcefulness training includes teaching self-help (stress-management, problem-solving) and help-seeking skills, respectively. Biofeedback training consists of the use of a hand-held device that shows the participant their changes in heart rate based on changes in their breathing pattern (as they relax); caregivers who need or prefer the biofeedback will be given a device to use for 28 days. All study participants receiving the intervention will also be asked to keep a journal to record their experience with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Have a living family member or a recently deceased family member diagnosed with Alzheimer's disease or another dementia
* Identify self as a primary caregiver
* In-home Caregivers: must be currently providing a minimum of 4 hours per day of supervision/direct care, and have entered that role within the past twelve months; Care Partners whose family member moved into a nursing or assisted living facility within the past twelve months, and must report visiting their care recipient at least once per week; Caretakers (i.e. bereaved) whose family member is deceased within the past twelve months, and are persons with direct oversight of the deceased person's belongings, estate, finances, etc.
* Be capable of performing informed consent and participating in study procedures

Exclusion Criteria:

* Does not have a family member with Alzheimer's disease or another dementia
* Has not cared for a living family member with dementia within the last 12 months, or the family member has been deceased for more than 12 months
* Has knowledge of another family member in the same household enrolled in the study
* Currently pregnant
* Has a pacemaker
* Lives outside of the study area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaclene A Zauszniewski, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- CWRU School of Nursing, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Family carers of elders with dementia will be recruited using various strategies (community support organizations, publicly posted flyers, online ads) in NE Ohio. Eligible participants were adults over the age of 18, who were carers of a family member (over the age of 65) with a medical diagnosis of dementia, and had transitioned to a new phase of caring in the previous 6 months.
Pre-assignment Details: Enrolled participants may be excluded if they elect not to participate after enrolling.
Groups:
- Need: Participants will be assigned to either Resourcefulness Training or HRV-focused Biofeedback interventions based on their need (as determined by baseline data).
  Resourcefulness Training: A cognitive-behavioral intervention presented within an audiovisual format that consists of teaching and reinforcing personal (self-help) and social (help-seeking) resourcefulness skills.
  Biofeedback Training: Use of a heart-rate variability (HRV) tracking device to enable one to learn to alter physiology to improve health. Devices are used to measure physiological activity, e.g., breathing and heart function, and provide rapid, accurate "feedback" to the user, thereby enabling desired physiological changes that can endure over time without continued use of the device and to continue to influence behavior.
- Preference: Participants will be given a choice of Resourcefulness Training or HRV-focused Biofeedback interventions.
  Resourcefulness Training: A cognitive-behavioral intervention presented within an audiovisual format that consists of teaching and reinforcing personal (self-help) and social (help-seeking) resourcefulness skills.
  Biofeedback Training: Use of a heart-rate variability (HRV) tracking device to enable one to learn to alter physiology to improve health. Devices are used to measure physiological activity, e.g., breathing and heart function, and provide rapid, accurate "feedback" to the user, thereby enabling desired physiological changes that can endure over time without continued use of the device and to continue to influence behavior.
- Attention Control: Participants assigned to the attention control group will be presented with Diversionary activities.
  Diversional Activites: An audiovisual format presenting 12 activities for adults including but not limited; crossword puzzles, reading, gardening, exercise, cooking/baking, board games, learning a new language, social activities, online games, etc.
Period: Overall Study
Arm/Group | Need | Preference | Attention Control
Started | 105 | 100 | 103
Completed | 90 | 85 | 88
Not Completed | 15 | 15 | 15
Not completed — Lost to Follow-up | 15 | 15 | 15

BASELINE CHARACTERISTICS:
Population: All participants who consented and completed the baseline questionnaire.
Groups:
- Need; Preference: Participants in this arm were, at enrollment, caregivers (in the home), care partners (with a care facility), or caretakers (bereaved) of persons with dementia. Those in this randomly assigned group were given a choice to participate in one of two self-management interventions (either biofeedback or resourcefulness training).
- Attention Control: Participants in this arm were, at enrollment, caregivers (in the home), care partners (with a care facility), or caretakers (bereaved) of persons with dementia. Those in this randomly assigned group participated in diversional activities.
- Total: Total of all reporting groups
Arm/Group | Need | Preference | Attention Control | Total
Number analyzed (Participants) | 105 | 100 | 103 | 308
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 10 | 9 | 30
  Between 18 and 65 years | 56 | 52 | 55 | 163
  >=65 years | 38 | 38 | 39 | 115
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 87 | 88 | 266
  Male | 14 | 13 | 15 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 2 | 5
  Not Hispanic or Latino | 105 | 97 | 101 | 303
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 20 | 12 | 16 | 48
  White | 82 | 84 | 85 | 251
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 105 | 100 | 103 | 308

OUTCOME MEASURES:

1. Primary Outcome: Change in Caregiver's Perceived Stress Scale
Description: 14 items; 3-point scale; Scores range 9-27; higher score indicates greater perceived stress
Time Frame: From T1 (baseline) to T2 (6 months) through T3 (one year)
Population: The overall analyzed participants included all who completed the T3 questionnaire across the three arms. 15 participants in each arm discontinued their participation between baseline (T1) and T3. Thus, this number equals 308 (who completed baseline measures) minus 45 (who dropped out over time) which equals 263 at T3.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Need | Preference | Attention Control
Number analyzed (Participants) | 90 | 85 | 88
score on a scale
  Baseline | 19.73 (7.97) | 21.01 (6.37) | 19.84 (7.48)
  T2 (6 months post baseline) | 19.21 (6.19) | 17.34 (6.97) | 16.95 (7.34)
  T3 (1 year post baseline) | 16.49 (6.55) | 18.40 (7.41) | 17.19 (7.54)

2. Primary Outcome: Change in Caregiver's Negative Emotions Checklist
Description: 10 items; dichotomous list; Scores range 0-10; higher score indicates more negative emotions.
Time Frame: From T1 (baseline) to T2 (6 months) through T3 (one year)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Need | Preference | Attention Control
Number analyzed (Participants) | 90 | 85 | 88
score on a scale
  Baseline | 6.80 (3.03) | 7.19 (2.55) | 6.19 (2.85)
  T2 (6 months post baseline) | 5.98 (3.12) | 5.97 (2.79) | 5.74 (3.04)
  T3 (1 year post baseline) | 5.47 (3.21) | 6.15 (2.97) | 6.06 (3.20)

3. Primary Outcome: Change in Caregiver's Depressive Cognitions Scales
Description: 8 items; 6-point scale; Scores range 0-40; higher score indicates higher depressive cognition
Time Frame: From T1 (baseline) to T2 (6 months) through T3 (one year)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Need | Preference | Attention Control
Number analyzed (Participants) | 90 | 85 | 88
score on a scale
  Baseline | 8.48 (6.36) | 10.22 (6.93) | 8.74 (7.09)
  T2 (6 months post baseline) | 10.00 (8.29) | 7.33 (6.13) | 7.4 (5.62)
  T3 (1 year post baseline) | 8.11 (6.78) | 8.96 (7.80) | 8.03 (5.96)

4. Primary Outcome: Change in Global Health - Physical Health: PROMIS (Patient Reported Outcomes Measurement Information System)
Description: Change in self-assessment of general physical health, as measured by the Patient-Reported Outcomes Measurement Information System 10-Question Short Form (PROMIS-10 Global Health). Ten items are rated on a five-point scale, scores range from 0-20, and a higher score indicates better health and health-related quality of life.
Time Frame: From T1 (baseline) to T2 (6 months) through T3 (one year)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Self-management Intervention Based on Need: Participants randomly assigned to this arm receive a self-management intervention (Resourcefulness Training or Biofeedback) according to baseline data.
  Resourcefulness training
  Biofeedback
- Self-management Intervention Based on Preference: Participants randomly assigned to this arm receive a self-management intervention (Resourcefulness Training or Biofeedback) according to their preference.
  Resourcefulness training
  Biofeedback
Arm/Group | Self-management Intervention Based on Need | Self-management Intervention Based on Preference | Attention Control: Diversonal Activities
Number analyzed (Participants) | 90 | 85 | 88
score on a scale
  Baseline | 14.80 (2.50) | 14.23 (2.39) | 14.10 (2.92)
  T2 (6 months post baseline) | 14.29 (4.94) | 14.67 (2.61) | 14.68 (2.77)
  T3 (1 year post baseline) | 14.75 (2.69) | 14.20 (2.64) | 14.31 (2.54)

5. Primary Outcome: Change in Caregiver Global Health - Mental Health: PROMIS (Patient Reported Outcomes Measurement Information System)
Description: Change in self-assessment of general mental health, as measured by the Patient-Reported Outcomes Measurement Information System 10-Question Short Form (PROMIS-10 Global Health). Ten items are rated on a five-point scale, scores range from 0-20, and a higher score indicates better health and health-related quality of life.
Time Frame: From T1 (baseline) to T2 (6 months) through T3 (one year)
Population: All participants who completed the T3 questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Need | Preference | Attention Control
Number analyzed (Participants) | 90 | 85 | 88
score on a scale
  Baseline | 12.31 (3.29) | 11.57 (2.95) | 12.44 (3.30)
  T2 (6 months post baseline) | 12.56 (3.05) | 12.90 (3.28) | 13.06 (3.18)
  T3 (1 year post baseline) | 13.01 (3.08) | 12.1 (3.27) | 12.86 (3.10)

6. Primary Outcome: Change in Caregiver's Health Risk Behavior Scale
Description: Measure of Caregiving Health Risks: 9 items; 3-point scale, Scores range 9-27; higher score indicates greater risk
Time Frame: From T1 (baseline) to T2 (6 months) through T3 (one year)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Need | Preference | Attention Control
Number analyzed (Participants) | 90 | 85 | 88
score on a scale
  Baseline | 15.97 (3.27) | 16.67 (3.77) | 16.19 (3.62)
  T2 (6 months post baseline) | 15.89 (3.09) | 15.54 (3.80) | 15.10 (3.12)
  T3 (1 year post baseline) | 15.24 (3.10) | 15.45 (3.52) | 15.17 (3.34)

ADVERSE EVENTS:
Time Frame: Data was collected for the duration of the study (one year post-baseline questionnaire).
Description: All events would have been reported. No adverse events occurred.
Arm/Group | Need | Preference | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/100 | 0/103
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/100 | 0/103
Other Adverse Events (participants affected / at risk) | 0/105 | 0/100 | 0/103

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT04603482/Prot_SAP_000.pdf